CLINICAL TRIAL: NCT01702337
Title: Additional Health and Economic Impact of the Bivalent Versus the Quadrivalent HPV Vaccine in Taiwan: Results of a Prevalence-based Model
Brief Title: Prevalence-based Health and Economic Model of the Bivalent Versus the Quadrivalent Human Papillomavirus (HPV) Vaccine
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114420
Record Dates: First submitted 2012-09-27; First posted 2012-10-08 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Human Papillomavirus Infection
Keywords: Gardasil; Prevalence-model; Cervarix; economic; health
MeSH Terms: conditions — Papillomavirus Infections

GROUPS / COHORTS (2):
- HPV-1 Group: Hypothetical group of women vaccinated with HPV-1 vaccine in Taiwan.
  Interventions: Other: Prevalence-based model
- HPV-2 Group: Hypothetical group of women vaccinated with HPV-2 vaccine in Taiwan.
  Interventions: Other: Prevalence-based model

INTERVENTIONS:
Other: Prevalence-based model — Static prevalence-based model to estimate vaccine effect over a one-year period at a steady state (when all women are fully vaccinated).

SUMMARY:
This study compares the health and economic impact of the bivalent HPV vaccine (HPV-1) and the quadrivalent HPV vaccine (HPV-2).

DETAILED DESCRIPTION:
This study uses a prevalence-based model (by using efficacy data from each vaccine's respective trials and published cost data for Taiwan) which estimates the differences in lesions, genital warts, cervical cancer and costs from a healthcare payer's perspective prevented between HPV-1 and HPV-2 vaccines during one year (when all women are vaccinated). It also analyses costs from a societal perspective.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects vaccinated with either HPV-1 or HPV-2 vaccines in Taiwan (hypothetical group).

Exclusion Criteria:

* Not applicable.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hypothetical group of women vaccinated with either HPV-1 or HPV-2 vaccines in Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Annual number of lesions prevented by each vaccine | Over a one-year period
Lesion related total cost averted by each vaccine | Over a one-year period
Additional costs averted by HPV-1 vaccine compared to HPV-2 vaccine | Over a one-year period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] ADDITIONAL HEALTH AND ECONOMIC IMPACT OF THE BIVALENT VERSUS THE QUADRIVALENT HPV VACCINE IN TAIWAN: RESULTS OF A PREVALENCE-BASED MODEL, Ho. T.H., van Enckevort, P.J. & Demarteau, N. Poster presented at: ISPOR, 4th Asia-Pacific Conference, 5-7 September 2010, Phuket, Thailand.